CLINICAL TRIAL: NCT01081652
Title: An Open, Randomized, Comparative, Phase III Study Using Micronised Progesterone (Crinone® 8%) in the Luteal Phase Support of Women Undergoing in Vitro Fertilization and Embryo Transfer (IVF/ET)
Brief Title: A Study Using Micronised Progesterone (Crinone® 8%) in the Luteal Phase Support of Women Undergoing in Vitro Fertilisation (IVF) and Embryo Transfer (ET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Medical Director, Serono Singapore, an affiliate of Merck KGaA, Darmstadt, Germany.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25347
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2010-03

CONDITIONS: Infertility
Keywords: Fertilisation, In vitro; Embryo transfer; progesterone; Reproductive technologies, Assisted
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — Progesterone

ARMS (2):
- Crinone 8% group (Experimental): Female subjects undergoing IVF/ET treated with Crinone 8% intravaginally
  Interventions: Drug: Micronised Progesterone
- Intramuscular progesterone group (Active Comparator): Female subjects undergoing IVF/ET treated with 60 mg progesterone intramuscularly once daily
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Micronised Progesterone — Micronised progesterone administered intravaginally once daily from the day of ET. If pregnancy was confirmed on day 14 of progesterone administration, progesterone was continued for another 45 days.
  Other Names: Crinone 8%
  Arms: Crinone 8% group
Drug: Progesterone — Progesterone 60 mg administered intramuscular once daily from the day of ET. If pregnancy was confirmed on day 14 of progesterone administration, progesterone was continued for another 45 days.
  Arms: Intramuscular progesterone group

SUMMARY:
This was an open-label, randomized, comparative, phase III study to evaluate the safety and efficacy of Crinone 8% in comparison with progesterone 60 mg intramuscular (i.m.) administered once a day in luteal phase support in 200 Chinese female subjects undergoing IVF/ET.

DETAILED DESCRIPTION:
This was an open-label, randomized, comparative, multicentric, phase III study to evaluate the safety and efficacy of Crinone 8% in comparison with progesterone 60 mg intramuscular administered once a day in luteal phase support in Chinese female subjects undergoing IVF/ET. The study planned to enroll 200 female subjects who underwent pituitary down-regulation as per each center's normal practice prior to and during stimulation of multiple follicular development. The progesterone administration was started on the day of ET. Randomisation was performed on the day of ET. If pregnancy was confirmed on day 14 of the progesterone administration, the progesterone was continued for another 45 days. The subjects were followed up and the treatment outcome (negative pregnancy test or pregnancy) was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent
* BMI < 25 kg/m2
* Age < 36 years
* <3 prior ART cycles (IVF, ICSI and related procedures)
* Infertility
* Regular spontaneous ovulatory menstrual cycles

Exclusion Criteria:

* Habitual abortion
* Hydrosalpinges
* History of past poor response to COH
* Patients with serious arterial, lung, hepatic and renal diseases
* Hepatic and renal impairment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2004-05; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The difference in hCG positive rate in the two arms 14 days after embryo transfer
The difference in pregnancy rates in the two arms 30 and 60 days after embryo transfer
The difference in implantation rate in the two arms 30 days after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Huafei Li, Study Director — Serono Pharmaceutical Limited
Locations (1):
- Peking University 3rd Hopistal, Beijing, China